CLINICAL TRIAL: NCT02379117
Title: Eating Behaviour in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 15005
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Crohn's Disease Patients: Patients with a diagnosis of Crohn's disease fitting the studies inclusion & exclusion criteria.
- Healthy Volunteers: For healthy volunteers the studies exclusion criteria apply.

SUMMARY:
Food intake is mainly controlled through interactions between the gut and brain (the homeostatic control) and through our environment, with food exposure, mood and past experiences (the hedonic control) playing a major role. The link between the gut and the brain is mainly controlled through enteroendocrine cells (EC). These cells in the bowel sense nutrients in the food and link with the brain to control how much we eat. They make a number of hormones that link with the brain to control one's eating habits.

Crohn's disease (CD) is an inflammatory disease of the bowel which can present with a number of symptoms including weight loss and loss of appetite. We thought some time ago that an increase in the number and function of these EC could play a central role. Since then we have carried out work which has shown that in CD these EC increase in number and produce more hormones after a meal. This finding could have a negative effect on food intake. This would be one explanation to the symptoms so commonly experienced by these patients.

In CD we thus feel that there might be an imbalance in the appetite control. We expect an increasingly sensitive gut to food intake and a subdued mood and perception to food reward and that this imbalance will lead to a decrease in food reward and consequently a decrease in food intake.

This study will be carried out using Healthy Volunteers and CD patients. We plan to measure food intake though telephone interviews and plan to analyse eating behaviour through 5 questionnaires.This study will help us to improve our understanding of what it is that controls food intake. This will be particularly important to patients with CD who routinely lose weight and appetite.

DETAILED DESCRIPTION:
STUDY BACKGROUND INFORMATION AND RATIONALE

Crohn's disease (CD) patients can present with a variety of luminal and extra-luminal symptoms but nutritional abnormalities are a very common but poorly studied [1] problem in this disease [2]. Apart from disease burden and repeated surgery, reduced appetite [3] and associated symptoms such as nausea undoubtedly contribute, with a major impact on quality of life.

Appetite and satiation, the processes by which a meal is terminated, involve complex interactions of homeostatic and hedonic factors. While the hypothalamus is central in the homeostatic control of food intake, other neural circuits integrate environmental and emotional cues to constitute the hedonic drive of appetite regulation. The homeostatic control of food intake is governed by the enteroendocrine-gut brain axis. Enteroendocrine cells (EC) play a pivotal role in orchestrating physiological functions in the gastrointestinal (GI) tract. Sensing the nutrient content of the lumen, they secrete multiple peptides and amines that control gut secretory and motor functions. Gut hormones act on vagal afferents in the GI tract, directly relaying to key central nervous system (CNS) nuclei that interface within the hypothalamus and other cortical areas to regulate food intake. CD patients with active small bowel inflammation show significant up-regulation of EC cells with an increase in ileal expression of chromogranin A [4, 5], glucagon-like peptide-1 (GLP-1) [4], key transcription factors in the stem cell to EC differentiation pathway [4] , plasma polypeptide YY (PYY) [3], cholecystokinin (CCK) [6] levels and a reduction in the key enzyme dipeptidyl peptidase-4 expression [7]. This increase in plasma peptide levels is associated with the symptoms of nausea and anorexia, with both symptoms, and tissue and plasma EC-peptide expression decreasing to normality in remission [3].

An increase in EC expression at the tissue and plasma level might affect appetite regulation through an increase in CNS signalling.

Fatty-acids infused in the gut, lead to a CCK-dependent increase in CNS activity in areas related to homeostatic control of feeding such as the brainstem, the pons, hypothalamus, cerebellum and the motor cortical areas [8]. Glucose has been shown to decrease the response in the upper hypothalamus [9], possibly via a GLP-1-mediated pathway [10]. Ghrelin and PYY have known homeostatic CNS signalling properties but play a hedonic role in the control of food intake [11]. In effect, the increase in plasma PYY and GLP-1 seen after Roux-en-Y gastric bypass surgery in obese subjects or after parenteral administration [12] is associated with a lower activation in brain-hedonic food responses and a healthier eating behaviour [13]. In CD, we expect a subdued reward value of food, but postulate that this would be aversive, and inappropriately impairing appetite and food intake.

We hypothesize that in CD and small bowel inflammation we will observe a change in eating behaviour with loss of hedonic drives and food reward responses and an accentuated homeostatic response.

STUDY OBJECTIVES AND PURPOSE

PURPOSE The overall purpose of the study is to quantify food intake in patients with active Crohn's disease and compare it to when they are in remission and to healthy age, BMI and gender-matched healthy cohort of volunteers. We will quantify eating behaviour traits in the same patient cohort when in active disease and repeat when in remission. These data will be compared to that of healthy volunteers.

PRIMARY OBJECTIVE The primary objective is to quantify food intake in patients with active CD and compare this to HV.

SECONDARY OBJECTIVES The secondary objectives of this study are to a) quantify food intake in patients with active CD and compare that when in inactive disease. b) quantify changes in appetite and eating behaviour in patients with active CD and compare these to those in HV and inactive CD as measured by the appetite-related questionnaires

ELIGIBILITY:
Inclusion Criteria:

-

We will study a cohort of CD patients with active disease as defined by:

1. Age 16-75 years
2. Ulceration seen at ileocolonoscopy, aiming for a simple endoscopic score for Crohn's disease (SES-CD) of 4-19, in the absence of stricturing disease or,
3. Intestinal inflammation or deep ulceration seen on CT or MR enterography, with the disease activity quantified via the MaRIA score or
4. Faecal calprotectin of >250µg/g or
5. C-Reactive protein >5mg/dl or,
6. Harvey-Bradshaw index score of 5-16
7. Body mass index (BMI) of 18-30.

For HV participants, inclusion criteria's 1 and 7 apply.

Exclusion Criteria:

1. Present or recent (within 12 weeks) corticosteroid usage
2. Malignant disease
3. BMI <18 or >30.
4. Significant cardiovascular or respiratory disease
5. Diabetes mellitus
6. Current Infection
7. Neurological or cognitive impairment; significant physical disability
8. Significant hepatic disease or renal failure
9. Abnormal blood results other than those explained by CD including bleeding diatheses (apart from in the case of HV where all unexplained blood results are an exclusion criteria) ,
10. Subjects currently participating in (or in the last three months) any other research project
11. pregnancy or breastfeeding or
12. Severe CD where a delay in a change in medical treatment for 1 weeks would not be clinically advisable

For HV participants, all exclusion criteria apply with the exception of criteria no.12

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment
  The chief investigator is a specialist in Inflammatory Bowel disease and also an associate professor of gastroenterology at the University of Nottingham and Nottingham University Hospital which is a tertiary-level care academic institution covering a population of approximately 1 million people for secondary-level care and 4.5 million people for tertiary-level care. Collectively we manage approximately 4000 IBD patients.
  Participants shall be recruited from two sources:
  1. Crohn's Disease patients from clinic.
  2. Crohns Disease patients and Healthy Volunteers via the study flyer and social media.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-04; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon W Moran, Principal Investigator — University of Nottingham
Locations (1):
- Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Result] Bryant RV, Trott MJ, Bartholomeusz FD, Andrews JM. Systematic review: body composition in adults with inflammatory bowel disease. Aliment Pharmacol Ther. 2013 Aug;38(3):213-25. doi: 10.1111/apt.12372. Epub 2013 Jun 14. PMID 23763279
- [Result] Lochs H, Dejong C, Hammarqvist F, Hebuterne X, Leon-Sanz M, Schutz T, van Gemert W, van Gossum A, Valentini L; DGEM (German Society for Nutritional Medicine); Lubke H, Bischoff S, Engelmann N, Thul P; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Gastroenterology. Clin Nutr. 2006 Apr;25(2):260-74. doi: 10.1016/j.clnu.2006.01.007. Epub 2006 May 15. PMID 16698129
- [Result] Moran GW, Leslie FC, McLaughlin JT. Crohn's disease affecting the small bowel is associated with reduced appetite and elevated levels of circulating gut peptides. Clin Nutr. 2013 Jun;32(3):404-11. doi: 10.1016/j.clnu.2012.08.024. Epub 2012 Sep 3. PMID 22999064
- [Result] Moran GW, Pennock J, McLaughlin JT. Enteroendocrine cells in terminal ileal Crohn's disease. J Crohns Colitis. 2012 Oct;6(9):871-80. doi: 10.1016/j.crohns.2012.01.013. Epub 2012 Mar 3. PMID 22398079
- [Result] Moran GW, McLaughlin JT. Plasma chromogranin A in patients with inflammatory bowel disease: a possible explanation. Inflamm Bowel Dis. 2010 Jun;16(6):914-5. doi: 10.1002/ibd.21096. No abstract available. PMID 19760780
- [Result] Keller J, Beglinger C, Holst JJ, Andresen V, Layer P. Mechanisms of gastric emptying disturbances in chronic and acute inflammation of the distal gastrointestinal tract. Am J Physiol Gastrointest Liver Physiol. 2009 Nov;297(5):G861-8. doi: 10.1152/ajpgi.00145.2009. PMID 20501434
- [Result] Moran GW, O'Neill C, Padfield P, McLaughlin JT. Dipeptidyl peptidase-4 expression is reduced in Crohn's disease. Regul Pept. 2012 Aug 20;177(1-3):40-5. doi: 10.1016/j.regpep.2012.04.006. Epub 2012 May 2. PMID 22561447
- [Result] Lassman DJ, McKie S, Gregory LJ, Lal S, D'Amato M, Steele I, Varro A, Dockray GJ, Williams SC, Thompson DG. Defining the role of cholecystokinin in the lipid-induced human brain activation matrix. Gastroenterology. 2010 Apr;138(4):1514-24. doi: 10.1053/j.gastro.2009.12.060. Epub 2010 Jan 18. PMID 20080096
- [Result] Smeets PA, de Graaf C, Stafleu A, van Osch MJ, van der Grond J. Functional magnetic resonance imaging of human hypothalamic responses to sweet taste and calories. Am J Clin Nutr. 2005 Nov;82(5):1011-6. doi: 10.1093/ajcn/82.5.1011. PMID 16280432
- [Result] Pannacciulli N, Le DS, Salbe AD, Chen K, Reiman EM, Tataranni PA, Krakoff J. Postprandial glucagon-like peptide-1 (GLP-1) response is positively associated with changes in neuronal activity of brain areas implicated in satiety and food intake regulation in humans. Neuroimage. 2007 Apr 1;35(2):511-7. doi: 10.1016/j.neuroimage.2006.12.035. Epub 2007 Jan 18. PMID 17317222
- [Result] Batterham RL, ffytche DH, Rosenthal JM, Zelaya FO, Barker GJ, Withers DJ, Williams SC. PYY modulation of cortical and hypothalamic brain areas predicts feeding behaviour in humans. Nature. 2007 Nov 1;450(7166):106-9. doi: 10.1038/nature06212. Epub 2007 Oct 14. PMID 17934448
- [Result] De Silva A, Salem V, Long CJ, Makwana A, Newbould RD, Rabiner EA, Ghatei MA, Bloom SR, Matthews PM, Beaver JD, Dhillo WS. The gut hormones PYY 3-36 and GLP-1 7-36 amide reduce food intake and modulate brain activity in appetite centers in humans. Cell Metab. 2011 Nov 2;14(5):700-6. doi: 10.1016/j.cmet.2011.09.010. Epub 2011 Oct 13. PMID 22000927
- [Result] Scholtz S, Miras AD, Chhina N, Prechtl CG, Sleeth ML, Daud NM, Ismail NA, Durighel G, Ahmed AR, Olbers T, Vincent RP, Alaghband-Zadeh J, Ghatei MA, Waldman AD, Frost GS, Bell JD, le Roux CW, Goldstone AP. Obese patients after gastric bypass surgery have lower brain-hedonic responses to food than after gastric banding. Gut. 2014 Jun;63(6):891-902. doi: 10.1136/gutjnl-2013-305008. Epub 2013 Aug 20. PMID 23964100

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crohn's Disease Patients | Healthy Volunteers
Started | 30 | 31
Completed | 30 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crohn's Disease Patients | Healthy Volunteers | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 31 | 60
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Inter-Quartile Range); unit: years] — years
  years | 32.3 [23 to 36.5] | 32.8 [25.5 to 35.5] | 32.5 [24 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 18 | 19 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Dietary Recalls (Calorific Intake)
Description: The primary endpoints for this study will be food intake as measured by one telephone-administered 24-h dietary recall. Total calorific intake will be calculated.
Time Frame: Participants will be included in this study for 1 week
Measure: Mean (Standard Error); unit: kcal
Arm/Group | Crohn's Disease Patients | Healthy Volunteers
Number analyzed (Participants) | 30 | 31
kcal | 1900.9 (138.6) | 2054.3 (110.7)

2. Secondary Outcome: Three Factor Eating Questionnaire (TFEQ) Restraint, Disinhibition and Hunger Subscales
Description: The TFEQ contains 51 items and measures three dimensions of human eating behaviour: Cognitive Restraint of Eating [I], Disinhibition [II], and Hunger [III]. Each item scores either 0 or 1 point. The minimum score for factors I, II. and III is therefore 0, with the pos- sible maximum scores being 21, 16, and 14 respectively. High scores mean worse outcome.
Time Frame: Healthy volunteer participants will be included in this study for 1 week. Crohn's Disease participants will be included in the study until they are re-assessed in remission. A time limit of 12 months will be given.
Reporting Status: Not Posted

3. Secondary Outcome: The Binge Eating Scale
Description: The BES is a 16-item questionnaire that assesses the severity of binge eating tendencies. Eight questions describe the behavioural mani- festations of binge eating behaviour and eight describe the feelings and cognitions associated with binge eating. Scores are summed to produce a total score ranging from 0 to 46. Cut-off points have previously been reported denoting mild [≤17], moderate [18-26], and severe [≥27] binge eating behaviours. High score means worse outcome
Time Frame: as for outcome 2
Reporting Status: Not Posted

4. Secondary Outcome: The Power of Food Scale
Description: The PFS is a 15-item questionnaire reflecting the psychological influence of the food environment. It measures appetite for, rather than consumption of, palatable foods and may be a useful measure of the hedonic impact of food environments replete with highly palatable foods. Items are grouped into three domains according to food proximity; food available but not physically present; food present but not tasted; and food tasted but not consumed. High scores mean worse outcome
Time Frame: as for outcome 2
Reporting Status: Not Posted

5. Secondary Outcome: The Dutch Eating Behaviour Questionnaire
Description: The 33-item DEBQ assesses different eating styles that may contribute to weight gain: emotional eating, external eating, and restraint. 'Emotional eating' occurs in response to emotional arousal states such as fear, anger, or anxiety; 'external eating' occurs in response to external food cues such as sight and smell of food; and 'restraint eating' is overeating after a period of slimming when the cognitive resolve to diet is abandoned. High score means worse outcome
Time Frame: as for outcome 2
Reporting Status: Not Posted

6. Secondary Outcome: The Control of Eating Questionnaire
Description: The CoEQ is a 21-item questionnaire designed to assess the severity and type of food cravings experienced over the previous 7 days. The CoEQ has four subscales: Craving Control, Craving for Savoury, Craving for Sweet, and Positive Mood. Items on the CoEQ are assessed by 100-mm visual analogue scales [VAS], with items relating to each subscale being averaged to create a final score. High positive mood is better outcome
Time Frame: as for outcome 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years 7 months
Description: Observational study, Cross sectional study, adverse events not monitored/assessed
Arm/Group | Crohn's Disease Patients | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT02379117/Prot_SAP_000.pdf